CLINICAL TRIAL: NCT04716101
Title: Ultrasound Imaging Measurements of the Thoracolumbar Fascia Following Massage Therapy: a Proof of Concept Study
Brief Title: Ultrasound Imaging Measurements of the Thoracolumbar Fascia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CE 19.358
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: Fascia; Quantitative ultrasound; Elastography; Massage therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with nonspecific low back pain (Experimental): Patients will be randomized to receive either a massage technique or a sham massage technique.
  Interventions: Other: Massage therapy technique; Other: Sham massage technique
- Asymptomatic volunteers (Active Comparator): Similarly, the volunteers will be randomized to receive either a massage technique or a sham massage technique.
  Interventions: Other: Massage therapy technique; Other: Sham massage technique

INTERVENTIONS:
Other: Massage therapy technique — The massage therapy technique consists of manual deep and slow compression and shearing forces applied on the lumbar spine muscles and thoracolumbar fascia in a distal to proximal direction.
Other: Sham massage technique — For the sham massage technique the massage therapist will put the right palm at the participant's right lower back along erector spinae and likewise left palm at left lower back without applying force, holding the palm during 2 minutes and half.

SUMMARY:
In this prospective study, eligible subjects with chronic non specific low back pain and asymptomatic volunteers will undergo a research dynamic ultrasound exam of the lower back before and after a massage technique.

The overall aim of the present research is to develop ultrasonographic parameters that characterize the geometrical, the mechanical and tissue characteristic properties of the thoracolumbar fascia, and to explore the effect of a massage therapy technique on these parameters.

DETAILED DESCRIPTION:
In this prospective proof of concept study, eligible subjects with chronic non specific low back pain and asymptomatic volunteers will undergo a research dynamic ultrasound (US) exam of the thoracolumbar fascia (TLF) of the lower back. A musculoskeletal radiologist will perform the US exams consisting of a series of 5 dynamic scans of both the right and left paraspinal muscles, obtained during 15 degrees of passive flexion of the lower body using a motorized table.

Following the US exam, the group of patients and the group of volunteers will be respectively randomized to receive either a standardized massage technique intervention or a sham technique. The US exam will be repeated after the intervention.

Ultrasound image segmentation will be performed by two independent observers and inter-rater variability will be assessed. Post-processing of the US recordings will include assessment of geometrical (thickness), mechanical (percent shear strain between the TLF and the epimysium-muscle complex) and tissue ultrastructure features (the mean intensity μ, the scatterer clustering parameter α and the structure parameter κ of the echo envelope). These features will be compared between patients and volunteers and between the intervention groups.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Presenting with chronic low back and/or referred pain (non specific pattern) above or just below the gluteal fold of at least 3/10 on a numerical pain rating scale (NRS), for at least 6 months;
* Pain is present at least 50% of the time during the day;

Asymptomatic group:

* No history of low back pain or any other chronic pain limiting activities of daily living or work.

Exclusion Criteria:

* History of back surgery;
* History of severe back or low extremity injury;
* Back pain attributable to a specific, recognizable, known pathology (i.e.: infection, tumor, fracture, spinal stenosis, sciatica etc.);
* Corticosteroid medication intake or corticosteroid injection in the lumbar spine in the previous 3 months;
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Shear Strain After the Massage Intervention | Baseline and immediately after the massage intervention.
  Percent shear strain between the thoracolumbar fascia and the epimysium of the erector spinae muscle.

SECONDARY OUTCOMES:
Thickness | Baseline
  Thickness (millimeters) of the thoracolumbar fascia.
Change from Baseline Quantitative Ultrasound Marker 'μ' After the Massage Intervention. | Baseline and immediately after the massage intervention.
  Statistical analysis of the echo envelope: the mean intensity μ. This marker is unitless.
Change from Baseline Quantitative Ultrasound Marker 'α' After the Massage Intervention. | Baseline and immediately after the massage intervention.
  Statistical analysis of the echo envelope: the scatterer clustering parameter α. This marker is unitless.
Change from Baseline Quantitative Ultrasound Marker 'κ' After the Massage Intervention. | Baseline and immediately after the massage intervention.
  Statistical analysis of the echo envelope: the structure parameter κ. This marker is unitless.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie J Bureau, MD MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tomita N, Roy-Cardinal MH, Chayer B, Daher S, Attiya A, Boulanger A, Gaudreault N, Cloutier G, Bureau NJ. Thoracolumbar fascia ultrasound shear strain differs between low back pain and asymptomatic individuals: expanding the evidence. Insights Imaging. 2025 Jan 15;16(1):18. doi: 10.1186/s13244-024-01895-2. PMID 39812963
- [Derived] Tomita N, Destrempes F, Cardinal MR, Boulanger A, Gaudreault N, Cloutier G, Bureau NJ. Thoracolumbar Fascia Microstructure and Low Back Pain: Insights From Quantitative Ultrasound Homodyned K-Distribution Statistical Modeling. Ultrasound Med Biol. 2025 Nov;51(11):2113-2119. doi: 10.1016/j.ultrasmedbio.2025.07.031. Epub 2025 Aug 23. PMID 40850900